CLINICAL TRIAL: NCT04790578
Title: Technology to Support Exercise Adherence in Project EXCEL Participants
Brief Title: EXCEL: Technology and Exercise Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREBA.CC-20-0283
Record Dates: First submitted 2021-03-01; First posted 2021-03-10 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: Exercise; mHealth
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants of the EXCEL study will be randomly allocated to either receiving the ZoeInsigths application during their 12 week baseline class + 12 week follow-up (intervention) or only receiving the 12 week baseline class (waitlist control). Those in the waitlist control group will be offered the ZoeInsights application at the end of the 24-week study period after completing their 24-week measures. Block randomization will be used so that all EXCEL participants in a single group-based class will be assigned to either the intervention or waitlist control group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be unaware of the intervention the participants received. Due to the nature of the intervention (a eHealth application) participants can't be blinded to the intervention. Furthermore, due to the intention to integrate the application as part of extended support provided in the EXCEL program, exercise class instructors (care providers) will be made aware of participant group assignment. The research coordinator will also be aware of the intervention of each participant to aid in troubleshooting with the ZoeInsights application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZoeInsights Application Arm (Experimental): Participants will receive free access to the ZI app for the 12-week intervention. After completing initial set-up, participants will be asked to record physical activity and symptoms regularly via scheduled in-app routines. Further use of ZI (eg. Custom daily routines, additional graphing, medication tracking, accessing linked health resources) during the intervention will be possible ad libitum. After the initial 12-weeks of the EXCEL+ZI intervention, participants have continued free access to the ZI app for up to 1 year.
  Interventions: Device: ZoeInsights Application; Behavioral: EXCEL Exercise Class
- Waitlist control (Active Comparator): During the 12-week intervention the participants will only take part in an online delivered EXCEL exercise class and will not have access to the ZI app. After completion of the 24-week test, the participants will be granted access to the ZI app.
  Interventions: Behavioral: EXCEL Exercise Class

INTERVENTIONS:
Device: ZoeInsights Application — ZI is designed to promote PA behavior change and maintenance via self-monitoring of PA, symptoms, and other health data. Additional information for using ZI will be provided via a PDF-based user guide on installing and using the application, a live instructional webinar hosted by ZI developer Hanalytics Solutions, and access to continued support via email/telephone communication with study staff as well as Hanalytics Solutions. Reminders to complete self-monitoring tasks will be provided using daily push notifications scheduled according to participant preferences. Automatic graphs will be generated and displayed within the app to allow participants to visualize trends in physical activity, symptoms, and other health data. ZI can be accessed via a web browser on any device that is connected to the internet (e.g. computer, laptop, tablet, smartphone), or via a native android or iOS mobile application on a smartphone or tablet.
  Arms: ZoeInsights Application Arm
Behavioral: EXCEL Exercise Class — The group based remote exercise program is delivered twice a week over the Zoom application. Classes are one hour long with a ten minute warm up, 40 minute strength and conditioning focused exercise circuits, and a ten minute stretching. Each class is followed by additional time to provide participants with an opportunity to interact with each other, fostering social support.

SUMMARY:
Exercise adherence and maintenance in the EXCEL program supported with a smart phone application: A pilot randomized controlled trial

DETAILED DESCRIPTION:
Purpose: The primary aim of this proposed pilot randomized controlled trial is to investigate the effectiveness and patterns of use of a mHealth application (ZoeInsights - ZI) for supporting physical activity (PA) maintenance in remote and rural cancer survivors within an online-delivered exercise oncology program (Project EXCEL; ethics HREBA-CC.20-0098).

Background/Rationale: Evidence indicates mixed effectiveness for online-delivered exercise oncology programs to improve physical activity (PA) behavior, especially with regards to maintenance of PA behavior post-intervention. Supportive resources are needed, especially for remote/rural cancer survivors who may have lower social support, PA self-efficacy, motivation, as well as unique barriers to PA. Mobile health technology (mHealth) has potential to support PA behavior change in cancer survivors, but evidence for its impact and best implementation practices in exercise oncology remains limited. Prior findings on PA behavior change suggest that in order to elicit lasting effects, early integration of supportive resources (eg. self-monitoring via a mhealth app) within PA participation is important. And in particular, research is needed to determine the effectiveness of mHealth within exercise oncology programs for supporting long-term PA maintenance. No studies on mhealth exercise interventions have been carried out in remote/rural cancer survivors.

Objectives: Primary aim is to assess the effectiveness of the mhealth app, ZI for supporting maintenance of PA behavior change, up to 24-weeks from program initiation. The impact of the ZI intervention on PA behaviour change will be measured by weekly objectively measured minutes of moderate to vigorous physical activity (MVPA), subjectively reported weekly minutes of MVPA, and program attendance. The investigators hypothesize the ZI intervention group will have improved maintenance of PA behavior change at 24-weeks compared to those in EXCEL only group. The secondary outcomes aim to assess the extent of use of the application. This will be assessed by app usage, satisfaction reports, and the participants perspectives on the continued use of the ZI application. The investigators hypothesize that majority of users will download and continue to use the application throughout the 24-week study period.

Methods:

Participants and Recruitment All EXCEL participants will be eligible to participate in the proposed sub-study, including those who may already be using PA-related apps. Email invitations will be sent to eligible participants with a study overview, instructions on who to contact to answer questions, and a link to complete the informed consent form in the EXCEL RedCap database if they are interested in participating. The consent form will require an electronic signature. It will be marked as complete in RedCap as soon as all required fields are completed and the participant submits the form. After completion of recruitment, randomization using a random number generator, with odd numbers assigned to the intervention (EXCEL + ZI at baseline) and even numbers to the waitlist control (EXCEL + ZI at 24 weeks) group. Randomization will occur by clusters so that all participants in the same exercise class day and time will be assigned to the intervention or waitlist control group. This will be done to enhance the integration of ZoeInsights within the EXCEL program.

To participate in EXCEL, participants must 1) have a cancer diagnosis; 2) be over the age of 18 years; 3) be able to participate in mild levels of activity as a minimum (to be assessed during screening via the Physical Activity Readiness Questionnaire); 4) be pre-treatment, or receiving active cancer treatment, or have received cancer treatment within the past three years; 5) be able to provide informed written consent in English; and 6) have access to internet service that can support video calling. All EXCEL participants live in rural or remote locations in Canada. The inclusion criteria ensures the investigators reach a wide range of cancer survivors throughout various stages of their journey while ensuring they are physically capable of safely completing exercise. Participants will be eligible regardless of cancer type and stage and there are no aims to recruit specific cancer survivors. No stratification for treatment status will occur.

Study Design/Procedure The proposed study will be a prospective, 2-arm, pilot randomized controlled trial with waitlist control arm. Participants randomized to the intervention will receive access to the ZI application for the duration of the study. Those in the waitlist control group will be able to download and use ZI after completing the 24-week assessment. All participants will take part in the standard 12-week group-based EXCEL online exercise program. Garmin wearable PA trackers will be provided to all participants to objectively track PA habits throughout the intervention.

Intervention

The ZI App:

ZI is designed to promote PA behavior change and maintenance via self-monitoring of physical activity, symptoms, and other health data. Furthermore, self-monitoring is intended to facilitate participant understanding of and communication about their PA and health with caregivers, exercise professionals, and healthcare professionals. Additional information for using ZI will be provided via a PDF-based user guide on installing and using the application, a live instructional webinar hosted by ZI developer Hanalytics Solutions, and access to continued support via email/telephone communication with study staff as well as Hanalytics Solutions. After completing initial set-up, participants will be asked to record physical activity and symptoms regularly via scheduled in-app routines. Reminders to complete these self-monitoring tasks will be provided using daily push notifications scheduled according to participant preferences. Automatic graphs will be generated and displayed within the app to allow participants to visualize trends in physical activity, symptoms, and other health data. Further use of ZI (eg. Custom daily routines, additional graphing, medication tracking, accessing linked health resources) during the intervention will be possible ad libitum.

ZI can be accessed via a web browser on any device that is connected to the internet (e.g. computer, laptop, tablet, smartphone), or via a native android or iOS mobile application on a smartphone or tablet. No devices will be provided to participants, as participants are already required to own an internet-connected device for email communication and completion of study measures online in RedCap.

The EXCEL online exercise program:

The EXCEL exercise program is based on the Alberta Cancer Exercise (ACE) program (HREBA.CC-16-0905), adapted as required for rural/remote site implementation. The exercise program includes a combination of aerobic, resistance, balance, and flexibility exercises delivered in a circuit-type class setting or group personal training format, twice weekly for a 8-12 week period. The exercise sessions will be conducted online in small groups of 8-15 participants under the direct supervision of a trained qualified exercise professional (QEP). The sessions will be conducted over the Zoom platform and the QEP will be provided additional support from the central research team, including moderators for sessions. The exercises will be slightly modified to ensure safety of all participants is maintained, based on current ACE online delivery. The program follows exercise progression principles (ie, principles of frequency, intensity, time, type, overload and progression) over the 8-12-weeks, with tailoring of any exercise to meet individual participant needs as required, in order to promote fitness and wellness benefits.

Timing Participants will complete the baseline assessment, including EXCEL and sub-study-specific questionnaires and baseline physical function assessment, prior to EXCEL class start (T0). They will then be given access, within the first two weeks of EXCEL, to the ZI application along with the ZI user guide and invitation to the instructional webinar to facilitate installation, set-up, and familiarization with ZI. Upon program start, participants will attend twice-weekly group-based EXCEL exercise classes and use ZI as outlined above to self-monitor PA and health. The study will consist of 2 phases, the intervention phase (EXCEL classes + ZI) from week 0-12, followed by the maintenance phase from weeks 12-24 (ZI only). Outcome measures will be collected at 3 subsequent time points: week 4 (T1), week 12 (T2), and week 24 (T3).

Measures Demographics (T0) Participant demographics will be collected within EXCEL. Additionally, participants will be asked to complete a set of questionnaires to assess prior technology usage, familiarity, and literacy.

Physical Activity (T0-T3) To examine effectiveness of ZI to support PA habits and maintenance, PA will be assessed via self-report at all time points (T0-T3) using the Godin Leisure Time Exercise Questionnaire (GLTEQ) and objectively throughout the intervention using the accelerometer (continued reporting of objective PA via Garmin after T2 is optional). In addition, class attendance (weeks 1-12) will be recorded.

Patterns of ZI use (T1-T3) App usage data will be collected directly via ZI, including logins, tasks completed, pages visited, additional use, and continued usage habits during the maintenance phase. User satisfaction with ZI as well as usability will be assessed using the validated mobile app usability questionnaire (MAUQ). Additional data collected includes error reporting/technical difficulties and costs of providing ZI per participant (subscription fee and support hours required). Participant perceptions of using the ZI application will be examined via qualitative semi-structured interviews.

Qualitative Interviews (T2-T3) A purposive sample of participants from the intervention group (n=10-20) will be invited to participate in semi-structured one-on-one interviews at 12 and 24 weeks. Interviews will focus on participant perspectives of using the ZI app as well as its usefulness for supporting PA behavior change and maintenance. An interview guide was developed by researchers with open-ended questions that are designed to guide the discussion while allowing the participant voice to dictate the flow of their interview. Purposive sampling will be used to ensure that participants from various demographic backgrounds are represented, giving consideration to age, gender, cancer diagnosis (type, stage, time since diagnosis), and baseline technology use.

EXCEL Study Measures (T0, T2, T3) As part of the EXCEL study, participants will complete a online physical function assessment with a clinical exercise physiologist (CEP). The CEP will assess resting health measures (heart rate, blood pressure, height, weight) as well as measures of flexibility, strength, and endurance via standardized tests. EXCEL participants will also complete questionnaires assessing symptom burden (Edmonton Symptom Assessment Scale), quality of life (Functional Assessment of Cancer Therapy - General and Cognitive subscales), fatigue (Functional Assessment of Chronic Illness Therapy - Fatigue subscale), and exercise barriers and facilitators (Exercise Barriers and Facilitators questionnaire developed for ACE).

Sample Size The sample size calculation is based on the primary outcome of assessing intervention effectiveness for supporting PA maintenance. A total sample of 140 (70 per group) provides at least 80% power to detect a between-group difference in PA of 60 minutes per week (including any PA from mild housework to strenuous training) with a two-tailed alpha of 5%, allowing for 10% attrition over the intervention period. The investigators do not anticipate that the second wave of EXCEL (Winter 2020) will recruit more than 60-80 participants, thus the investigators will collect data over at least two waves. Preliminary analyses on feasibility, and any changes required, would be made at the end of Spring 2021 session (i.e., July 2021), and put into place for Fall 2021 participants.

Data Analysis Participant baseline characteristics and patterns of use will be summarized using descriptive statistics. To investigate within and between-group differences at all time points, random effects linear mixed models will be used. The models will be controlled for potential demographic confounders (age, gender, cancer type, treatment status, and others). Primary analyses will follow intention-to-treat principles, with exploratory subgroup analyses based on actual ZI usage (i.e. completion of routines and other self-monitoring). Qualitative interviews will be transcribed verbatim and analyzed according to interpretive description methodology based on a constructivist philosophy.

ELIGIBILITY:
Inclusion Criteria

* Have a cancer diagnosis
* Be over the age of 18 years
* Be able to participate in mild levels of activity as a minimum (to be assessed during screening via the Physical Activity Readiness Questionnaire)
* Be pre-treatment, or receiving active cancer treatment, or have received cancer treatment within the past three year
* Be able to provide informed written consent in English
* Have access to internet service that can support video calling
* Be signed up for the EXCEL baseline class

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Physical Activity Minutes Per Week | Measured continuously from baseline to 24 weeks
  Change in activity levels from pre to post; Number of participants meeting Guidelines for Physical Activity of 90 minutes per week of moderate to vigorous intensity exercise, based on accelerometer data from commercially-available activity tracker.
  For the activity tracker each minute in the 55-70 percent age predicted HRmax will be evaluated as moderate intensity and above 70 percent of HRmax will be evaluated as vigorous intensity.
  Vigorous intensity minutes of physical activity will be doubled and added with moderate intensity minutes to obtain moderate to vigorous physical activity (MVPA) minutes.
Subjective Physical Activity Minutes Per Week | Self-reported at baseline, week 4, week 12, and week 24
  Change in Physical Activity minutes per week, based on modified Godin Leisure Time Exercise Questionnaire (mGLTEQ). In the mGLTEQ all dimensions (strenuous exercise, moderate exercise, mild exercise, resistance training, and flexibility) will be looked at separately and weekly minutes will be calculated by multiplying duration times frequency of sessions. Vigorous intensity minutes of exercise will be doubled and added with moderate intensity minutes to obtain moderate to vigorous physical activity (MVPA) minutes. Higher scores are better, indicating more minutes of MVPA were accumulated.
EXCEL class attendance | Potential class data in EXCEL baseline and maintenance classes will be recorded, and input into REDCap, from week 1-12 (baseline); and 12-24 (maintenance, optional)
  Class attendance (up to 2 x per week) during weeks 1-12 will be recorded by the EXCEL class lead, and input into REDCap. In addition, attendance at subsequent EXCEL maintenance programs (up to week 24) will be recorded

SECONDARY OUTCOMES:
ZI application usage | Continuous measurement from baseline to 24 weeks
  Measured directly through the app as logins, tasks completed, pages visited, additional use, and continued usage habits during the maintenance phase
Participant Satisfaction | Completed at week 4, 12, and 24
  Change in the mobile app usability questionnaire (MAUQ) score. Scores for each item range from 0 (strongly disagree) to 7 (strongly agree), with higher scores indicating greater satisfaction.
Body Composition | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in body mass index (BMI)
Aerobic Endurance | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in 6-minute walk test (m) or 2 minute step test (steps) results
Upper extremity grip strength | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in hand-grip dynamometry (kg)
Functional performance test | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in sit-to-stand (number of repetitions in 30 seconds)
Upper extremity flexibility | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in active shoulder flexion range of motion (degrees)
Lower extremity flexibility | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in sit-and-reach test (cm)
Balance | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in one legged stance test (seconds)
Cancer related symptoms | Assessed at baseline and weeks 4, 8, 12, 16, 20, 24
  Change in Edmonton Symptom Assessment Scale. Scores range from 0 to 10 for each item, with a total score ranging from 0 to 100. Higher scores indicate higher symptom burden.
General Health-related Quality of Life | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in EuroQual - 5 Dimensions (EQ-5D) tool. Scores for each item range from 1 to 5, with lower scores indicating better quality of life.
Fatigue | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in Functional Assessment of Chronic Illness Therapy - Fatigue subscale
  - scale is from 0-4, where 0 means "not at all" and 4 means "very much".
General well-being | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in Functional Assessment of Cancer Therapy - General subscale
  - scale is from 0-4, where 0 means "not at all" and 4 means "very much".
Cognition | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in Functional Assessment of Cancer Therapy - Cognitive subscale
  - scale is from 0-4, where 0 means "never" and 4 means "several times a day" (experiencing symptoms).
Barriers and facilitators to exercise participation | Assessed at baseline,12-weeks (post-intervention), and 24 weeks (follow-up)
  Change in Exercise Barriers and Facilitators questionnaire
Exercise adherence | Continuous measurement from baseline to 24 weeks
  Adherence to exercise programming (attendance at sessions)
Participant perceptions of using the ZI application | At 12 and 24 weeks
  A purposive sample of participants from the intervention group (n=10-20) will be invited to participate in semi-structured one-on-one interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Ester M, Wagoner CW, Dreger J, Chen G, McDonough MH, McNeely ML, Culos-Reed SN. Effectiveness of a Self-Monitoring App in Supporting Physical Activity Maintenance Among Rural Canadians With Cancer After an Exercise Oncology Program: Cluster Randomized Controlled Trial. JMIR Cancer. 2023 Sep 7;9:e47187. doi: 10.2196/47187. PMID 37676714